CLINICAL TRIAL: NCT00428870
Title: Arthroscopic Decompression Versus Diagnostic Arthroscopy Without Subacromial Decompression Versus Supervised Exercise Therapy in Treatment of Subacromial Impingement Syndrome. A Blinded Randomized Controlled Trail.
Brief Title: Operative or Conservative Treatment for Subacromial Impingement Syndrome?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Mika Paavola, MD, PhD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R04200
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Shoulder; impingement; conservative; acromioplasty; arthroscopy
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Arthroscopy; salicylhydroxamic acid; Conservative Treatment; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Arthroscopic acromioplasty (Experimental): Arthroscopic acromioplasty
  Interventions: Procedure: Arthroscopic acromioplasty or arthroscopy alone (sham) or conservative treatment (rehabilitation)
- Sham surgery (Placebo Comparator): Shoulder arthroscopy without active treatment and subacromial arthroscopy without bursectomy, decompression or other active interventions
  Interventions: Procedure: Arthroscopic acromioplasty or arthroscopy alone (sham) or conservative treatment (rehabilitation)
- Conservative treatment (Active Comparator): Standardized exercise rehabilitation (supervised by physiotherapist)
  Interventions: Procedure: Arthroscopic acromioplasty or arthroscopy alone (sham) or conservative treatment (rehabilitation)

INTERVENTIONS:
Procedure: Arthroscopic acromioplasty or arthroscopy alone (sham) or conservative treatment (rehabilitation)

SUMMARY:
pShoulder impingement syndrome is common and number of operations done per year is growing. The aim of this study is to compare the value of arthroscopic subacromial decompression (acromioplasty group) vs. diagnostic arthroscopy (control group) vs. supervised exercise therapy (conservative group) on subjects with chronic subacromial impingement syndrome. The results of treatment are measured at 3 months, 6 months, 12 months, 24 months, 5 years and 10 years. Primary outcome measures are pain at rest and activity (VASs) and secondary outcomes are functional assessment of the shoulder with Constant score and Simple Shoulder test (SST), global assessment of change , quality of life assessment (SF-36 and 15D) and costs. At 10 year follow-up, MRI imaging is obtained and the findings compared to baseline imaging.

DETAILED DESCRIPTION:
Applicant information:

Name: Mika Paavola, MD, PhD Address: Helsinki University Central Hospital, Töölö Hospital, Topeliuksenkatu 5, P.O. Box 266, FIN-00029 HUS, Finland Tel: +358 50 523 8382 Fax: +358 9 471 87481 Email: mika.paavola@hus.fi

Trial record details:

Protocol / serial number: N/A Title: Arthroscopic decompression versus diagnostic arthroscopy without subacromial decompression versus supervised exercise therapy in treatment of subacromial impingement syndrome. A blinded randomized controlled trail.

Acronym: N/A Study hypothesis: Operative and diagnostic arthroscopy is equally effective as conservative treatment (supervised exercise therapy) alone for subacromial impingement syndrome.

Research ethics review: Ethics committee approval from the Ethics Committee of the Hospital Districts of Pirkanmaa, date 28.12.2004 (ETL code R04200) Study design: Randomized controlled trial

Participants - inclusion criteria: In the first phase orthopaedists select consecutive female or male patients who are admitted to the hospital policlinic of Helsinki University Hospital, (either Töölö Hospital or Jorvi Hospital) or District Hospital of Tampere (Hatanpää Hospital) and fulfill the following inclusion criteria:

1. Subjects are 35 to 65 years of age female or male and have a characteristic history and symptoms of subacromial impingement syndrome at least 3 months.
2. Symptoms have no relieved with appropriate conservative treatment (i.e. physiotherapy, NSAIDs and subacromial corticosteroid injection).
3. They have clinical findings of impingement syndrome; painful arc sign and pain in shoulder abduction, positive findings in two of three isometric shoulder abduction tests (0 degree, 30 degree and external rotation), and positive subacromial injection test.

Participants - exclusion criteria:

1. Previous surgery of affected shoulder
2. Symptomatic osteoarthrosis of acromio-clavicular joint
3. Full thickness rotator cuff tear based on clinical findings and MRI
4. Long-term cervical syndrome
5. Instability of shoulder
6. Reluctance to participate in any study groups (i.e. any treatment options of the study)
7. Reduced co-operation (drug or alcohol abuse, mental illness) Anticipated start date: 1/10/2005 Anticipated end date: 31/12/2009 Target number of participants: 210 Disease: Chronic (> 3 months before inclusion) shoulder subacromial pain syndrome.

Interventions: The aim of this study is to compare the value of arthroscopic subacromial decompression (acromioplasty group) vs. diagnostic arthroscopy (control group) vs. supervised exercise therapy (conservative group) on subjects with chronic subacromial impingement syndrome. The shoulder arthroscopy is done three to six week after the baseline clinical examination by one of the seven experienced shoulder orthopaedists. At first, arthroscopy of shoulder joint is performed in patients of acromioplasty group and control group, and all pathological findings are recorded. Thereafter, arthroscopy of subacromial space is carried out. In control group, subacromial decompression is not done. In patients of supervised exercised therapy group, 3 months period of exercise therapy with home exercises, supervised by experienced physiotherapist, is initiated.

Primary outcome(s): Pain at rest and activity assessed with 10-cm visual analog scales (VASs). Participants assess maximum pain in the previous two days at rest and at exertion. Main follow-up time-point is 24 months after initiation of the treatment (i.e. operative treatment or first visit at the physiotherapist. Other time-points when the main outcome is measured are before the randomization, three month follow-up, six month follow-up and 12 month follow-up.

Secondary outcome(s): Functional assessment of the shoulder with Constant score and Simple Shoulder test (SST), global assessment of change [symptom questionnaire and subjective contentment (10-cm visual analog scales)], quality of life assessment (SF-36 and 15D).

Sources of funding: Finnish Office for Health Technology Assessment (National Research and Development Centre for Welfare and Health of Finland) and Sigrid Juselius Foundation Main sponsor information Name: Finnish Office for Health Technology Assessment Address: National Research and Development Centre for Welfare and Health (STAKES) - P.O. Box 220, FI-00531 Helsinki, Lintulahdenkuja 4, Finland Contact person

Contact information:

Name: Mika Paavola Address: Department of Orthopedics and Traumatology, Töölö hospital, Helsinki University Central Hospital P.O. Box 266 00029 HUS Helsinki Finland Tel: +358-50-5238382 Email: mika.paavola@hus.fi and mika.paavola@fimnet.fi Privacy level: Show all contact details

ELIGIBILITY:
Inclusion Criteria:

In the first phase orthopaedists select consecutive female or male patients who are admitted to the hospital policlinic of Helsinki University Hospital, (either Töölö Hospital or Jorvi Hospital) or District Hospital of Tampere (Hatanpää Hospital) and fulfill the following inclusion criteria:

1. Subjects are 35 to 65 years of age female or male and have a characteristic history and symptoms of subacromial impingement syndrome at least 3 months.
2. Symptoms have no relieved with appropriate conservative treatment (i.e. physiotherapy, NSAIDs and subacromial corticosteroid injection).
3. They have clinical findings of impingement syndrome; painful arc sign and pain in shoulder abduction, positive findings in two of three isometric shoulder abduction tests (0 degree, 30 degree and external rotation), and positive subacromial injection test.

Exclusion Criteria:

1. Previous surgery of affected shoulder
2. Symptomatic osteoarthrosis of acromio-clavicular joint
3. Full thickness rotator cuff tear based on clinical findings and MRI
4. Long-term cervical syndrome
5. Instability of shoulder
6. Reluctance to participate in any study groups (i.e. any treatment options of the study)
7. Reduced co-operation (drug or alcohol abuse, mental illness)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2005-02; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pain at rest | 2 years (primary)
  Assessed with 10-cm visual analog scales (VASs).
Pain during activity | 2 years (primary)
  Assessed with 10-cm visual analog scales (VASs).

SECONDARY OUTCOMES:
Constant score and Simple Shoulder test | 2 years (primary)
  Functional assessment of the shoulder
global assessment of change, | 2 years (primary)
  Likert scale
SF-36 and 15D | 2 years (primary)
  Quality of life assessment
Costs | 2 years (primary)
  Resource use

CONTACTS AND LOCATIONS:
Overall Officials: Mika Paavola, MD, PhD, Principal Investigator — 1.1.2003; Teppo Jarvinen, MD, PhD, Study Chair — 1.1.2004; Antti Malmivaara, MD, PhD, Study Chair — 1.8.2004; Timo Järvelä, MD, PhD, Study Chair — 1.1.2004; Simo Taimela, MD, PhD, Study Chair — 1.6.2004; Harri Sintonen, Professor, Study Chair — 1.8.2004
Locations (1):
- Helsinki University Hospital, Töölö Hospital, Helsinki, HUS, Finland

REFERENCES:
- [Derived] Kanto K, Back M, Ibounig T, Bjorkenheim R, Malmivaara A, Czuba T, Inkinen J, Kalske J, Savolainen V, Sinisaari I, Toivonen P, Taimela S, Jarvinen TLN, Paavola M; Finnish Shoulder Impingement Arthroscopy Controlled Trial (FIMPACT) Investigators. Arthroscopic subacromial decompression versus placebo surgery for subacromial pain syndrome: 10 year follow-up of the FIMPACT randomised, placebo surgery controlled trial. BMJ. 2025 Dec 2;391:e086201. doi: 10.1136/bmj-2025-086201. PMID 41330610
- [Derived] Back M, Paavola M, Aronen P, Jarvinen TLN, Taimela S; Finnish Shoulder Impingement Arthroscopy Controlled Trial (FIMPACT) Investigators. Return to work after subacromial decompression, diagnostic arthroscopy, or exercise therapy for shoulder impingement: a randomised, placebo-surgery controlled FIMPACT clinical trial with five-year follow-up. BMC Musculoskelet Disord. 2021 Oct 19;22(1):889. doi: 10.1186/s12891-021-04768-7. PMID 34666734
- [Derived] Kanto K, Lahdeoja T, Paavola M, Aronen P, Jarvinen TLN, Jokihaara J, Ardern CL, Karjalainen TV, Taimela S. Minimal important difference and patient acceptable symptom state for pain, Constant-Murley score and Simple Shoulder Test in patients with subacromial pain syndrome. BMC Med Res Methodol. 2021 Mar 6;21(1):45. doi: 10.1186/s12874-021-01241-w. PMID 33676417
- [Derived] Paavola M, Malmivaara A, Taimela S, Kanto K, Inkinen J, Kalske J, Sinisaari I, Savolainen V, Ranstam J, Jarvinen TLN; Finnish Subacromial Impingement Arthroscopy Controlled Trial (FIMPACT) Investigators. Subacromial decompression versus diagnostic arthroscopy for shoulder impingement: randomised, placebo surgery controlled clinical trial. BMJ. 2018 Jul 19;362:k2860. doi: 10.1136/bmj.k2860. PMID 30026230
- [Derived] Paavola M, Malmivaara A, Taimela S, Kanto K, Jarvinen TL; FIMPACT Investigators. Finnish Subacromial Impingement Arthroscopy Controlled Trial (FIMPACT): a protocol for a randomised trial comparing arthroscopic subacromial decompression and diagnostic arthroscopy (placebo control), with an exercise therapy control, in the treatment of shoulder impingement syndrome. BMJ Open. 2017 Jun 6;7(5):e014087. doi: 10.1136/bmjopen-2016-014087. PMID 28588109